CLINICAL TRIAL: NCT05022563
Title: Treatment Patterns and Clinical Outcomes Among Venous Thromboembolism Patients Treated With Anticoagulants After the Entry of Non-vitamin K Antagonist Oral Anticoagulants in Korea
Brief Title: Treatment Patterns and Bleeding Risk of Anticoagulants in Patients With Venous Thromboembolism in Korea
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: X9001305; VTE HIRA Study (Other: Alias Study Number)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2022-09

CONDITIONS: Venous Thromboembolism
Keywords: Venous thromboembolism; anticoagulant; treatment pattern; bleed
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage | interventions — Warfarin; apixaban; Rivaroxaban; Dabigatran; edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (3):
- Parenteral anticoagulant only: LMWH, UFH
  Interventions: Drug: Parenteral anticoagulant
- Warfarin-based: Warfarin only + parenteral anticoagulant bridged warfarin
  Interventions: Drug: Warfarin
- NOAC-based: NOAC only + parenteral anticoagulant bridged NOAC
  NOAC: apixaban, rivaroxaban, dabigatran, edoxaban
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Dabigatran; Drug: Edoxaban

INTERVENTIONS:
Drug: Parenteral anticoagulant — Parenteral anticoagulant only
  Groups: Parenteral anticoagulant only
Drug: Warfarin — Warfarin-based
  Groups: Warfarin-based
Drug: Apixaban — Apixaban
  Groups: NOAC-based
Drug: Rivaroxaban — Rivaroxaban
  Groups: NOAC-based
Drug: Dabigatran — Dabigatran
  Groups: NOAC-based
Drug: Edoxaban — Edoxaban
  Groups: NOAC-based

SUMMARY:
This study is a retrospective, observational, nationwide population-based cohort study utilizing the South Korea's Health Insurance and Review Assessment Service (HIRA) database. The aims of this study are to describe the sociodemographic and clinical characteristics of patients with venous thromboembolism according to their anticoagulant treatment (parenteral anticoagulants, warfarin, or non-vitamin K antagonist oral anticoagulants), to describe the treatment patterns related to anticoagulants, and to examine the risk of major bleeding according to the specific type of oral anticoagulants. The study will be conducted in two phases: Phase I for descriptive study and Phase II for comparative study.

ELIGIBILITY:
Inclusion Criteria:

1. Incident VTE diagnosis in an inpatient or outpatient setting between 1 Mar 2013 and 30 Jun 2019
2. Received anticoagulation therapy (all medication codes for anticoagulants approved for VTE in Korea; UFH, LMWH, warfarin, and NOACs) within 30 days of their VTE diagnosis (the index date will be defined as the date of treatment initiation with anticoagulants)
3. Aged ≥18 years at index date

Exclusion Criteria:

1. Had a record of VTE diagnosis within the 12-month period prior to the index VTE encounter.
2. Diagnosed with atrial fibrillation/flutter, mechanical heart valve replacement or mitral stenosis anytime prior to index date
3. Had a record of Inferior Vena Cava filter anytime prior to index date
4. Received anticoagulatory therapy within the 12-month period prior to index VTE encounter
5. Prescribed two different anticoagulants on the same index date
6. Had a record of pregnancy within the 9-month period prior to index date
7. Had a record of active cancer within the past 6 months of period prior to index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with venous thromboembolism from the South Korea's Health Insurance Review and Assessment Service (HIRA) database between Mar 1, 2013 and Jun 30, 2019
Sampling Method: Probability Sample
Enrollment: 55759 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si
  - Sungkyunkwan University, Suwon

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=X9001305

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of participants diagnosed with venous thromboembolism (VTE) between 1 Mar 2013 and 30 Jun 2019 and received first prescription of anticoagulants within 30 days of VTE diagnosis in real world clinical practice, were retrieved from South Korea's health insurance review and assessment service (HIRA) database. Available data were extracted and evaluated during approximately 1 month of this retrospective observational study.
Pre-assignment Details: Study was to be conducted in 2 phases. Phase 1: to describe anticoagulant treatment pattern according to index VTE treatment (PAC only, warfarin based, NOAC based treatment). Phase 2: to compare risk of major bleeding according to specific type of OAC treatment. But, as assessed by real world data review committee Phase 2 was not conducted due to insufficient statistical power that would lead to small and imbalanced sample sizes in comparison groups. Only Phase 1 data were studied and reported.
Groups:
- Warfarin-Based Therapy: Participants diagnosed with VTE, initiated warfarin-based therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- Non-vitamin K Antagonist Oral Anticoagulants (NOAC)-Based Therapy: Apixaban: Participants diagnosed with VTE, initiated apixaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- NOAC-Based Therapy: Dabigatran: Participants diagnosed with VTE, initiated dabigatran (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- NOAC-Based Therapy: Edoxaban: Participants diagnosed with VTE, initiated edoxaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- NOAC-Based Therapy: Rivaroxaban: Participants diagnosed with VTE, initiated rivaroxaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- Parenteral Anticoagulants (PAC) Only: Participants diagnosed with VTE, initiated PAC only therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
Period: Overall Study
Arm/Group | Warfarin-Based Therapy | Non-vitamin K Antagonist Oral Anticoagulants (NOAC)-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | Parenteral Anticoagulants (PAC) Only
Started | 11208 | 5047 | 2103 | 2342 | 26276 | 8783
Without Active Cancer | 10390 | 4543 | 1894 | 2078 | 23049 | 6550
With Active Cancer (Diagnosis of Cancer Within Past 6 Months of Index Date) | 818 | 504 | 209 | 264 | 3227 | 2233
Completed | 11208 | 5047 | 2103 | 2342 | 26276 | 8783
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study.
Groups:
- NOAC-Based Therapy: Apixaban: Participants diagnosed with VTE, initiated apixaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- PAC Only: Participants diagnosed with VTE, initiated PAC only therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- Total: Total of all reporting groups
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only | Total
Number analyzed (Participants) | 11208 | 5047 | 2103 | 2342 | 26276 | 8783 | 55759
Age, Customized [Count of Participants; unit: Participants] — Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer: 18-40 years | 974 | 269 | 138 | 142 | 2042 | 527 | 4092
    Without Active Cancer: 40-65 years | 2920 | 998 | 481 | 479 | 6456 | 1643 | 12977
    Without Active Cancer: >=65 years | 6496 | 3276 | 1275 | 1457 | 14551 | 4380 | 31435
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer: 18-40 years | 7 | 2 | 4 | 4 | 68 | 59 | 144
    With Active Cancer: 40-65 years | 232 | 170 | 54 | 91 | 1007 | 927 | 2481
    With Active Cancer: >=65 years | 579 | 332 | 151 | 169 | 2152 | 1247 | 4630
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer: Female | 5978 | 2958 | 1126 | 1288 | 13498 | 3671 | 28519
    Without Active Cancer: Male | 4412 | 1585 | 768 | 790 | 9551 | 2879 | 19985
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer: Female | 394 | 256 | 101 | 117 | 1526 | 1095 | 3489
    With Active Cancer: Male | 424 | 248 | 108 | 147 | 1701 | 1138 | 3766
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of Participants According to Type of Index VTE Event [Count of Participants; unit: Participants] — Index VTE event included Deep Vein Thrombosis (DVT) only, and Pulmonary Embolism (PE) with or without DVT. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer: DVT only | 4232 | 2265 | 499 | 689 | 10919 | 2822 | 21426
    Without Active Cancer: PE with/without DVT | 6158 | 2278 | 1395 | 1389 | 12130 | 3728 | 27078
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer: DVT only | 264 | 164 | 44 | 71 | 918 | 735 | 2196
    With Active Cancer: PE with/without DVT | 554 | 340 | 165 | 193 | 2309 | 1498 | 5059
Number of Participants With Major Orthopedic Surgery-provoked VTE [Count of Participants; unit: Participants] — Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer | 183 | 78 | 53 | 43 | 480 | 119 | 956
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer | 2 | 2 | 1 | 1 | 10 | 6 | 22
Number of Participants According to Health Insurance Type [Count of Participants; unit: Participants] — In this baseline measure, number of participant with their health insurance type such as national health insurance, medical aid, and veterans were reported. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer: National Health Insurance | 9418 | 4156 | 1703 | 1889 | 21088 | 5845 | 44099
    Without Active Cancer: Medical aid | 969 | 387 | 191 | 188 | 1953 | 698 | 4386
    Without Active Cancer: Veterans | 3 | 0 | 0 | 1 | 8 | 7 | 19
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer: National Health Insurance | 748 | 471 | 195 | 240 | 3014 | 2123 | 6791
    With Active Cancer: Medical aid | 68 | 33 | 14 | 23 | 213 | 109 | 460
    With Active Cancer: Veterans | 2 | 0 | 0 | 1 | 0 | 1 | 4
Number of Participants Classified According to the Index Year [Count of Participants; unit: Participants] — In this baseline measure, number of participants were classified according to the index year in which they started receiving anticoagulants. Index year was defined as the year in which the treatment was initiated for the participants. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer: 2012 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Without Active Cancer: 2013 | 3035 | 0 | 4 | 0 | 1085 | 804 | 4928
    Without Active Cancer: 2014 | 2631 | 2 | 3 | 0 | 2994 | 955 | 6585
    Without Active Cancer: 2015 | 1664 | 224 | 345 | 0 | 4039 | 1012 | 7284
    Without Active Cancer: 2016 | 1188 | 837 | 540 | 182 | 4160 | 1118 | 8025
    Without Active Cancer: 2017 | 939 | 1144 | 547 | 537 | 4215 | 1116 | 8498
    Without Active Cancer: 2018 | 679 | 1496 | 304 | 825 | 4438 | 1021 | 8763
    Without Active Cancer: 2019 | 254 | 840 | 151 | 534 | 2118 | 524 | 4421
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer: 2012 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    With Active Cancer: 2013 | 253 | 0 | 0 | 0 | 165 | 244 | 662
    With Active Cancer: 2014 | 213 | 0 | 0 | 0 | 441 | 366 | 1020
    With Active Cancer: 2015 | 131 | 19 | 32 | 0 | 503 | 381 | 1066
    With Active Cancer: 2016 | 79 | 64 | 65 | 14 | 605 | 361 | 1188
    With Active Cancer: 2017 | 79 | 117 | 66 | 43 | 584 | 355 | 1244
    With Active Cancer: 2018 | 47 | 174 | 31 | 109 | 631 | 358 | 1350
    With Active Cancer: 2019 | 16 | 130 | 15 | 98 | 298 | 168 | 725
Charlson Comorbidity Index (CCI) [Mean (Standard Deviation); unit: Units on a scale] — CCI included myocardial infarction, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic pulmonary disease, rheumatologic disease, peptic ulcer disease, mild liver disease, moderate/severe liver disease, diabetes with and without chronic complication, hemiplegia or paraplegia, renal disease, any malignancy (including leukemia and lymphoma), metastatic solid tumor, and AIDS/HIV. CCI score range from 0 to 33, where "0" = low comorbid condition and "33" = high comorbid condition, higher scores indicated more comorbidity and higher mortality risk. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Units on a scale
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer | 1.21 (1.39) | 1.23 (1.37) | 1.21 (1.43) | 1.22 (1.38) | 1.15 (1.37) | 1.45 (1.61) | 1.22 (1.41)
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer | 4.84 (2.83) | 4.74 (2.85) | 4.77 (2.77) | 4.69 (2.95) | 5.02 (2.99) | 5.09 (3.00) | 4.98 (2.96)
HAS-BLED Score [Mean (Standard Deviation); unit: Units on a scale] — In this baseline measure, HAS-BLED score was assessed by combining score of 8 risk factors (hypertension, abnormal kidney function, abnormal liver function, age > 65 years, stroke, bleeding history, labile international normalized ratio [INR], and drugs [antiplatelet agents and Non-steroidal anti-inflammatory drugs {NSAIDs}] or alcohol use). Score ranged from 0-9, where "0" indicates low risk and "9" indicates high risk, where higher scores indicated more bleeding risk. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Units on a scale
    Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Without Active Cancer | 2.19 (1.16) | 2.31 (1.09) | 2.24 (1.10) | 2.24 (1.10) | 2.16 (1.11) | 2.26 (1.18) | 2.20 (1.13)
    With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    With Active Cancer | 2.45 (1.11) | 2.41 (1.07) | 2.46 (1.10) | 2.47 (1.14) | 2.38 (1.13) | 2.23 (1.17) | 2.35 (1.14)
Number of Participants With Previous use of Medications [Count of Participants; unit: Participants] — In this baseline measure, previous use of medications such as corticosteroids, non-steroidal anti-inflammatory drug (NSAIDs), angiotensin-converting-enzyme inhibitors (ACE) inhibitors, angiotensin II receptor blockers, anti-platelets, beta-blockers, calcium-channel blockers, selective serotonin reuptake inhibitors (SSRI), proton pump inhibitors, diuretics, thiazides, vasodilators, estrogens, cyclooxygenase-2 inhibitors, and triazole antifungal agents were reported. A participant could have used more than 1 medication. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Corticosteroids: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Corticosteroids: Without Active Cancer | 5109 | 1787 | 797 | 726 | 10415 | 2492 | 21326
    Corticosteroids: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Corticosteroids: With Active Cancer | 531 | 266 | 121 | 129 | 2066 | 1403 | 4516
    NSAIDs: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    NSAIDs: Without Active Cancer | 8135 | 3657 | 1492 | 1622 | 18695 | 4774 | 38375
    NSAIDs: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    NSAIDs: With Active Cancer | 670 | 397 | 172 | 225 | 2601 | 1704 | 5769
    ACE inhibitors: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    ACE inhibitors: Without Active Cancer | 4840 | 2086 | 867 | 1005 | 10036 | 3052 | 21886
    ACE inhibitors: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    ACE inhibitors: With Active Cancer | 513 | 295 | 122 | 160 | 1920 | 1163 | 4173
    Angiotensin II receptor blockers: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Angiotensin II receptor blockers: Without Active Cancer | 5083 | 2364 | 961 | 1108 | 10925 | 3283 | 23724
    Angiotensin II receptor blockers: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Angiotensin II receptor blockers: With Active Cancer | 397 | 233 | 103 | 130 | 1492 | 888 | 3243
    Antiplatelets: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Antiplatelets: Without Active Cancer | 3958 | 1763 | 752 | 868 | 8580 | 2773 | 18694
    Antiplatelets: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Antiplatelets: With Active Cancer | 229 | 159 | 58 | 84 | 895 | 507 | 1932
    Beta-blockers: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Beta-blockers: Without Active Cancer | 2124 | 825 | 361 | 432 | 4218 | 1272 | 9232
    Beta-blockers: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Beta-blockers: With Active Cancer | 155 | 72 | 44 | 53 | 547 | 293 | 1164
    Calcium-channel blockers: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Calcium-channel blockers: Without Active Cancer | 3522 | 1680 | 658 | 778 | 7703 | 2436 | 16777
    Calcium-channel blockers: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Calcium-channel blockers: With Active Cancer | 311 | 181 | 82 | 102 | 1161 | 698 | 2535
    SSRI: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    SSRI: Without Active Cancer | 725 | 404 | 170 | 216 | 1913 | 464 | 3892
    SSRI: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    SSRI: With Active Cancer | 41 | 28 | 17 | 17 | 190 | 98 | 391
    Proton pump inhibitors: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Proton pump inhibitors: Without Active Cancer | 2995 | 1607 | 693 | 759 | 7550 | 1925 | 15529
    Proton pump inhibitors: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Proton pump inhibitors: With Active Cancer | 398 | 262 | 112 | 152 | 1656 | 1057 | 3637
    Diuretics: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Diuretics: Without Active Cancer | 2270 | 796 | 379 | 425 | 4066 | 1306 | 9242
    Diuretics: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Diuretics: With Active Cancer | 337 | 183 | 78 | 113 | 1379 | 770 | 2860
    Thiazides: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Thiazides: Without Active Cancer | 2168 | 842 | 359 | 385 | 4253 | 1133 | 9140
    Thiazides: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Thiazides: With Active Cancer | 139 | 65 | 22 | 28 | 403 | 245 | 902
    Vasodilators: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Vasodilators: Without Active Cancer | 2532 | 1109 | 466 | 505 | 5595 | 1593 | 11800
    Vasodilators: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Vasodilators: With Active Cancer | 128 | 86 | 42 | 45 | 467 | 274 | 1042
    Estrogens: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Estrogens: Without Active Cancer | 182 | 96 | 21 | 43 | 466 | 108 | 916
    Estrogens: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Estrogens: With Active Cancer | 23 | 12 | 5 | 3 | 62 | 37 | 142
    Cyclooxygenase-2 inhibitors: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Cyclooxygenase-2 inhibitors: Without Active Cancer | 1184 | 1044 | 360 | 389 | 3956 | 929 | 7862
    Cyclooxygenase-2 inhibitors: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Cyclooxygenase-2 inhibitors: With Active Cancer | 72 | 70 | 29 | 26 | 332 | 216 | 745
    Triazole antifungal agents: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Triazole antifungal agents: Without Active Cancer | 774 | 329 | 130 | 129 | 1675 | 383 | 3420
    Triazole antifungal agents: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Triazole antifungal agents: With Active Cancer | 55 | 33 | 13 | 20 | 219 | 120 | 460
Number of Participants With Comorbidities [Count of Participants; unit: Participants] — In this baseline measure, number of participants with various comorbidities such as antiphospholipid syndrome, asthma, history of cancer, chronic obstructive pulmonary disease (COPD), chronic kidney disease, chronic liver disease, diabetes mellitus, fracture, heart failure, hyperlipidemia, hypertension, ischemic heart disease, myocardial infarction, stroke, and trauma were reported. A participant can have more than 1 comorbidity. Population: Baseline characteristic is reported in separate rows for participants with active cancer and without active cancer.
  Participants
    Antiphospholipid syndrome: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Antiphospholipid syndrome: Without Active Cancer | 280 | 85 | 42 | 41 | 589 | 76 | 1113
    Antiphospholipid syndrome: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Antiphospholipid syndrome: With Active Cancer | 8 | 8 | 1 | 4 | 91 | 87 | 199
    Asthma: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Asthma: Without Active Cancer | 1184 | 424 | 203 | 236 | 2351 | 546 | 4944
    Asthma: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Asthma: With Active Cancer | 92 | 44 | 26 | 23 | 271 | 152 | 608
    History of cancer: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    History of cancer: Without Active Cancer | 897 | 524 | 196 | 253 | 2432 | 904 | 5206
    History of cancer: With Active Cancer: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
    History of cancer: With Active Cancer |  |  |  |  |  |  | 0
    COPD: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    COPD: Without Active Cancer | 1766 | 707 | 332 | 370 | 3765 | 1010 | 7950
    COPD: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    COPD: With Active Cancer | 179 | 81 | 46 | 50 | 706 | 390 | 1452
    Chronic kidney disease: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Chronic kidney disease: Without Active Cancer | 312 | 87 | 32 | 45 | 294 | 215 | 985
    Chronic kidney disease: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Chronic kidney disease: With Active Cancer | 32 | 14 | 5 | 6 | 60 | 40 | 157
    Chronic liver disease: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Chronic liver disease: Without Active Cancer | 800 | 392 | 146 | 145 | 1723 | 537 | 3743
    Chronic liver disease: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Chronic liver disease: With Active Cancer | 91 | 68 | 28 | 37 | 456 | 339 | 1019
    Diabetes mellitus: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Diabetes mellitus: Without Active Cancer | 1818 | 866 | 326 | 335 | 3826 | 1454 | 8625
    Diabetes mellitus: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Diabetes mellitus: With Active Cancer | 161 | 92 | 51 | 65 | 695 | 455 | 1519
    Fracture: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Fracture: Without Active Cancer | 1137 | 511 | 258 | 273 | 2601 | 802 | 5582
    Fracture: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Fracture: With Active Cancer | 43 | 37 | 15 | 15 | 202 | 118 | 430
    Heart failure: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Heart failure: Without Active Cancer | 538 | 207 | 99 | 123 | 906 | 273 | 2146
    Heart failure: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Heart failure: With Active Cancer | 29 | 8 | 6 | 1 | 67 | 35 | 146
    Hyperlipidemia: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Hyperlipidemia: Without Active Cancer | 1735 | 1093 | 363 | 432 | 4452 | 1225 | 9300
    Hyperlipidemia: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Hyperlipidemia: With Active Cancer | 130 | 99 | 44 | 68 | 584 | 377 | 1302
    Hypertension: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Hypertension: Without Active Cancer | 4525 | 2086 | 821 | 920 | 9679 | 2916 | 20947
    Hypertension: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Hypertension: With Active Cancer | 335 | 205 | 79 | 97 | 1284 | 772 | 2772
    Ischemic heart disease: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Ischemic heart disease: Without Active Cancer | 235 | 91 | 34 | 60 | 463 | 201 | 1084
    Ischemic heart disease: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Ischemic heart disease: With Active Cancer | 15 | 10 | 3 | 8 | 60 | 25 | 121
    Myocardial infarction: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Myocardial infarction: Without Active Cancer | 53 | 25 | 10 | 6 | 88 | 89 | 271
    Myocardial infarction: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Myocardial infarction: With Active Cancer | 4 | 4 | 0 | 0 | 8 | 8 | 24
    Stroke: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Stroke: Without Active Cancer | 956 | 394 | 182 | 220 | 1987 | 796 | 4535
    Stroke: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Stroke: With Active Cancer | 56 | 27 | 17 | 15 | 172 | 96 | 383
    Trauma: Without Active Cancer: number analyzed (Participants) | 10390 | 4543 | 1894 | 2078 | 23049 | 6550 | 48504
    Trauma: Without Active Cancer | 43 | 10 | 4 | 4 | 67 | 20 | 148
    Trauma: With Active Cancer: number analyzed (Participants) | 818 | 504 | 209 | 264 | 3227 | 2233 | 7255
    Trauma: With Active Cancer | 1 | 1 | 0 | 0 | 8 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Interruption in Index Anticoagulant Treatment
Description: Treatment interruption was defined as when a participant had a gap with no new treatment within 30 days of the estimated end of supply of index treatment, but subsequently restarted the index treatment after this period of 30 days. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: From index date up to treatment interruption, during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: Analysis population included all eligible participants whose medical records were retrieved and observed in this study. 'NOAC-based therapy' arm considered all NOACs as one entity, while individual NOAC results discriminated between each NOAC, therefore total number of participants with outcome in NOAC-based therapy is not equal to sum of individual NOACs. Here, "Number Analyzed" signifies participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Groups:
- NOAC-Based Therapy: Participants diagnosed with VTE, initiated NOAC-based (apixaban, dabigatran, edoxaban, or rivaroxaban) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Participants
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 172 | 961 | 115 | 51 | 38 | 728 | 401

2. Primary Outcome: Time to Treatment Interruption
Description: Treatment interruption was defined as when a participant had a gap with no new treatment within 30 days of the estimated end of supply of index treatment, but subsequently restarted the index treatment after this period of 30 days. The time to treatment interruption was defined as the period from the index date to the date of treatment interruption. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: as for outcome 1
Population: All eligible participants whose medical records were retrieved and observed in this study. 'NOAC-based therapy' arm considered all NOACs as 1 entity, while individual NOAC results discriminated between each NOAC, hence total number of participants with outcome in NOAC-based therapy is not equal to sum of individual NOACs. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure with interruption event;"Number Analyzed": participants evaluable for specified rows.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 3601 | 9130 | 1080 | 543 | 477 | 6701 | 1627
Days
  Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Without Active Cancer | 163 [50 to 343] | 129 [37 to 189] | 86 [16 to 181] | 137 [56 to 188] | 130 [42 to 189] | 128 [38 to 188] | 3 [1 to 10]
  With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  With Active Cancer | 129 [50 to 270] | 137 [51 to 188] | 123 [59 to 186] | 119 [58 to 188] | 159 [30 to 199] | 134 [49 to 187] | 61 [7 to 160]

3. Primary Outcome: Number of Participants Who Switched to Another Anticoagulant Therapy
Description: Treatment switching was defined as a prescription of another anticoagulant therapy that was started after the treatment initiation of the index anticoagulant treatment and within 30 days after the estimated end of supply of the index anticoagulant drug (exposure to the new anticoagulant treatment must last for at least 30 days to be considered as a treatment switch). The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: From index date up to treatment switch, during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Participants
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 1541 | 1273 | 319 | 276 | 204 | 1777 | 535
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 144 | 173 | 33 | 30 | 26 | 208 | 208

4. Primary Outcome: Time to Treatment Switch
Description: Treatment switching was defined as a prescription of another anticoagulant therapy that was started after the treatment initiation of the index anticoagulant treatment and within 30 days after the estimated end of supply of the index anticoagulant drug (exposure to the new anticoagulant treatment must last for at least 30 days to be considered as a treatment switch). The time to treatment switch was defined as the period from the index date to the date of treatment switch. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: as for outcome 3
Population: All eligible participants whose medical records were retrieved and observed in this study. 'NOAC-based therapy' arm considered all NOACs as 1 entity, while individual NOAC results discriminated between each NOAC, hence total number of participants with outcome in NOAC-based therapy is not equal to sum of individual NOACs. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure with switch event; "Number Analyzed": participants evaluable for specified rows.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Days
  Without Active Cancer: number analyzed (Participants) | 1541 | 1273 | 319 | 276 | 204 | 1777 | 535
  Without Active Cancer | 57 [21 to 182] | 179 [53 to 199] | 66 [24 to 181] | 105 [32 to 189] | 87 [25 to 189] | 99 [23 to 189] | 27 [19 to 39]
  With Active Cancer: number analyzed (Participants) | 144 | 173 | 33 | 30 | 26 | 208 | 208
  With Active Cancer | 36 [13 to 99] | 76 [20 to 172] | 44 [14 to 109] | 60 [30 to 174] | 98 [28 to 150] | 53 [21 to 149] | 49 [27 to 102]

5. Primary Outcome: Number of Participants Who Completely Discontinued Index Anticoagulant Treatment
Description: Treatment discontinuation (complete discontinuation; no reinitiation) was defined as when a participant who ended their first continuous treatment episode with the index anticoagulant treatment without switching, and subsequently have no further prescriptions for that respective anticoagulant treatment during all available follow-up time. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: From index date up to treatment discontinuation, during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Participants
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449

6. Primary Outcome: Time to Treatment Discontinuation
Description: Treatment discontinuation (complete discontinuation; no reinitiation) was defined as when a participant who ended their first continuous treatment episode with the index anticoagulant treatment without switching, and subsequently have no further prescriptions for that respective anticoagulant treatment during all available follow-up time. The time to treatment discontinuation was defined as the period from the index date to the date of treatment discontinuation. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: as for outcome 5
Population: All eligible participants whose medical records were retrieved and observed in this study. 'NOAC-based therapy' arm considered all NOACs as 1 entity, while individual NOAC results discriminated between each NOAC,hence total number of participants with outcome in NOAC-based therapy is not equal to sum of individual NOACs. "Overall Number of Participants Analyzed":participants evaluable for this outcome measure with discontinuation event;"Number Analyzed":participants evaluable for specified rows.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 5151 | 22396 | 3107 | 1143 | 1311 | 16138 | 5983
Days
  Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Without Active Cancer | 129 [31 to 244] | 119 [34 to 185] | 84 [16 to 176] | 134 [60 to 186] | 154 [58 to 190] | 119 [31 to 185] | 2 [1 to 7]
  With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  With Active Cancer | 75 [26 to 184] | 101 [35 to 180] | 99 [35 to 179] | 118 [46 to 178] | 112 [44 to 187] | 97 [31 to 179] | 25 [4 to 95]

7. Primary Outcome: Overall Index Anticoagulant Treatment Duration
Description: Overall anticoagulant treatment duration was defined as the time period from the index date to the earliest of treatment interruption, switch, or discontinuation. Treatment interruption: when a participant had a gap with no new treatment within 30 days of estimated end of supply of index treatment, but subsequently restarted index treatment after this period of 30 days. Treatment switching: a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Treatment discontinuation: when a participant who ended their first continuous treatment episode with index anticoagulant treatment without switching, and subsequently have no further prescriptions for that respective anticoagulant treatment during all available follow-up time. The index date was defined as the date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: From index date up to the earliest of treatment interruption, switch, or discontinuation; during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- NOAC Based Therapy: Apixaban: Participants diagnosed with VTE, initiated apixaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- NOAC Based Therapy: Dabigatran: Participants diagnosed with VTE, initiated dabigatran (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
- NOAC Based Therapy: Edoxaban: Participants diagnosed with VTE, initiated edoxaban (NOAC-based) therapy in real world practice within 30 days of their VTE diagnosis between 1 March 2012 and 30 June 2019, were included in this cohort.
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC Based Therapy: Apixaban | NOAC Based Therapy: Dabigatran | NOAC Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Days
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 139 [36 to 317] | 140 [39 to 191] | 96 [21 to 185] | 137 [54 to 188] | 164 [58 to 202] | 128 [34 to 189] | 3 [1 to 12]
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 80 [25 to 192] | 111 [39 to 184] | 104 [42 to 182] | 105 [44 to 178] | 123 [41 to 198] | 102 [34 to 182] | 34 [7 to 115]

8. Primary Outcome: Number of Participants Who Were Persistent on Index Anticoagulant Treatment for 3 Months
Description: Participants were considered to be persistent on index anticoagulant treatment if a participant had evidence of a repeat prescription within 30 days of the end of their prescription and does not experience any of the events that included treatment interruption (participant had a gap with no new treatment within 30 days of estimated end of supply of index treatment, but subsequently restarted index treatment after 30 days), switch (prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug), or discontinuation (participant ended their first continuous treatment episode with index anticoagulant treatment without switching, and subsequently have no further prescriptions for that respective anticoagulant treatment during all available follow-up time). Index date: date of first prescription for anticoagulants within 30 days after the index VTE event.
Time Frame: Within 3 months of index date, during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC Based Therapy: Apixaban | NOAC Based Therapy: Dabigatran | NOAC Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Participants
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 6313 | 19848 | 2390 | 1225 | 1395 | 14037 | 222
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 388 | 2405 | 290 | 120 | 148 | 1770 | 673

9. Primary Outcome: Number of Participants Who Were Persistent on Index Anticoagulant Treatment for 6 Months
Description: as for outcome 8
Time Frame: Within 6 months of index date, during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 11208 | 35768 | 5047 | 2103 | 2342 | 26276 | 8783
Participants
  Without Active Cancer: number analyzed (Participants) | 10390 | 31564 | 4543 | 1894 | 2078 | 23049 | 6550
  Without Active Cancer | 4393 | 10557 | 1213 | 606 | 817 | 7209 | 75
  With Active Cancer: number analyzed (Participants) | 818 | 4204 | 504 | 209 | 264 | 3227 | 2233
  With Active Cancer | 217 | 1089 | 125 | 46 | 91 | 773 | 221

10. Primary Outcome: Number of Participants With Clinical Events Preceding Index Anticoagulant Treatment Interruption
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment interruption. Treatment interruption was defined as when a participant had a gap with no new treatment within 30 days of the estimated end of supply of index treatment, but subsequently restarted the index treatment after this period of 30 days. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event.
Time Frame: Within 30 days before treatment interruption during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 3601 | 9130 | 1080 | 543 | 477 | 6701 | 1627
Participants
  Major Bleeding: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Major Bleeding: Without Active Cancer | 27 | 53 | 5 | 2 | 2 | 42 | 4
  Complications of VTE: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Complications of VTE: Without Active Cancer | 6 | 13 | 0 | 3 | 0 | 10 | 5
  Thromboembolism: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Thromboembolism: Without Active Cancer | 158 | 328 | 50 | 19 | 18 | 233 | 209
  Major Surgery: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Major Surgery: Without Active Cancer | 92 | 566 | 126 | 9 | 17 | 407 | 171
  Cancer-related Event: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Cancer-related Event: Without Active Cancer | 62 | 126 | 14 | 5 | 4 | 99 | 100
  Kidney Function Changes: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Kidney Function Changes: Without Active Cancer | 45 | 87 | 10 | 8 | 7 | 55 | 44
  Liver Function Change: Without Active Cancer: number analyzed (Participants) | 3429 | 8169 | 965 | 492 | 439 | 5973 | 1226
  Liver Function Change: Without Active Cancer | 79 | 158 | 12 | 7 | 6 | 129 | 72
  Major Bleeding: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Major Bleeding: With Active Cancer | 1 | 8 | 3 | 0 | 0 | 4 | 2
  Complications of VTE: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Complications of VTE: With Active Cancer | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Thromboembolism: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Thromboembolism: With Active Cancer | 12 | 21 | 3 | 1 | 0 | 17 | 9
  Major Surgery: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Major Surgery: With Active Cancer | 15 | 33 | 1 | 2 | 1 | 27 | 55
  Cancer-related Event: With Active Cancer: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Kidney Function Changes: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Kidney Function Changes: With Active Cancer | 1 | 8 | 1 | 0 | 0 | 7 | 10
  Liver Function Change: With Active Cancer: number analyzed (Participants) | 172 | 961 | 115 | 51 | 38 | 728 | 401
  Liver Function Change: With Active Cancer | 2 | 9 | 3 | 1 | 0 | 5 | 9

11. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Major Bleeding
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "major bleeding" are reported.
Time Frame: Within 30 days before treatment switch during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: All eligible participants. 'NOAC-based therapy' arm considered all NOACs as 1 entity, while individual NOAC results discriminated between each NOAC, hence total number of participants with outcome in NOAC-based therapy is not equal to sum of individual NOACs. "Overall Number of Participants Analyzed": participants evaluable for this outcome measure with switch event. "Number Analyzed (n)": participants evaluable for specified rows. n =0 as switch in the same treatment arm not feasible.
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 5 | 0 | 0 | 1 | 4 | 5
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 17 |  |  |  |  |  | 11
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 0 | 1 | 0 | 0 | 0 | 1 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 2 |  |  | 1 | 1 | 9 | 1
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 3 |  | 0 |  | 0 | 2 | 1
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 0 |  | 3 | 0 |  | 3 | 2
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 12 |  | 0 | 1 | 0 |  | 7
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 1 | 0 | 0 | 0 | 1 | 0
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 0 |  |  |  |  |  | 0
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 0 | 1 | 0 | 0 | 0 | 1 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 0 |  |  | 0 | 0 | 1 | 0
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 0 |  | 0 |  | 0 | 0 | 0
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 0 |  | 0 | 0 |  | 2 | 0
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 0 |  | 0 | 0 | 0 |  | 0

12. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Complications of VTE
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "complications of VTE" are reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 12 | 0 | 0 | 0 | 11 | 1
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 2 |  |  |  |  |  | 2
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 0 | 0 | 0 | 0 | 0 | 0 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 0 |  |  | 0 | 0 | 1 | 0
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 1 |  | 0 |  | 0 | 0 | 0
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 0 |  | 1 | 0 |  | 2 | 0
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 0 |  | 0 | 0 | 0 |  | 2
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 0 | 0 | 0 | 0 | 0 | 0
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 0 |  |  |  |  |  | 0
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 0 | 0 | 0 | 0 | 0 | 0 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 0 |  |  | 0 | 0 | 0 | 0
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 0 |  | 0 |  | 0 | 0 | 0
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 0 |  | 0 | 0 |  | 0 | 0
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 0 |  | 0 | 0 | 0 |  | 0

13. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Thromboembolism
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "thromboembolism" are reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 59 | 6 | 3 | 2 | 48 | 12
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 108 |  |  |  |  |  | 51
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 5 | 15 | 1 | 0 | 1 | 13 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 8 |  |  | 1 | 4 | 30 | 6
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 9 |  | 1 |  | 3 | 15 | 3
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 7 |  | 9 | 1 |  | 25 | 6
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 85 |  | 14 | 6 | 9 |  | 36
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 9 | 1 | 0 | 0 | 8 | 4
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 12 |  |  |  |  |  | 8
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 7 | 9 | 0 | 0 | 1 | 8 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 1 |  |  | 0 | 0 | 4 | 1
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 3 |  | 0 |  | 0 | 1 | 1
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 0 |  | 1 | 0 |  | 1 | 1
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 8 |  | 0 | 3 | 0 |  | 5

14. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Major Surgery
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "major surgery" are reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 13 | 0 | 2 | 1 | 10 | 14
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 26 |  |  |  |  |  | 65
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 3 | 6 | 0 | 1 | 0 | 5 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 1 |  |  | 1 | 2 | 11 | 11
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 4 |  | 0 |  | 0 | 5 | 5
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 3 |  | 4 | 2 |  | 8 | 10
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 18 |  | 2 | 1 | 1 |  | 36
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 2 | 0 | 0 | 0 | 2 | 2
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 3 |  |  |  |  |  | 18
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 1 | 3 | 1 | 0 | 0 | 2 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 0 |  |  | 0 | 0 | 1 | 2
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 0 |  | 0 |  | 0 | 1 | 5
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 1 |  | 0 | 0 |  | 3 | 2
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 2 |  | 0 | 1 | 1 |  | 9

15. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Cancer-related Event
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "cancer-related event" are reported among participants without active cancer. Data not collected and reported for participants with active because all participants already had cancer.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1541 | 1273 | 319 | 276 | 204 | 1777 | 535
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 13 | 1 | 1 | 0 | 11 | 6
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 26 |  |  |  |  |  | 57
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 24 | 32 | 2 | 2 | 1 | 27 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 5 |  |  | 1 | 0 | 6 | 11
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 1 |  | 1 |  | 0 | 3 | 5
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 1 |  | 2 | 0 |  | 3 | 6
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 19 |  | 0 | 3 | 5 |  | 35

16. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Kidney Function Change
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "kidney function change" are reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 13 | 1 | 0 | 0 | 12 | 5
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 22 |  |  |  |  |  | 4
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 6 | 5 | 3 | 0 | 0 | 2 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 3 |  |  | 0 | 1 | 10 | 1
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 1 |  | 1 |  | 0 | 1 | 0
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 1 |  | 0 | 0 |  | 1 | 1
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 17 |  | 2 | 2 | 1 |  | 2
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 2 | 0 | 0 | 0 | 2 | 1
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 2 |  |  |  |  |  | 2
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 0 | 4 | 0 | 1 | 0 | 3 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 1 |  |  | 0 | 0 | 0 | 1
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 0 |  | 0 |  | 0 | 0 | 0
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 0 |  | 0 | 0 |  | 1 | 1
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 1 |  | 0 | 0 | 0 |  | 0

17. Primary Outcome: Number of Participants With Clinical Events Preceding Switch From Index Anticoagulant Treatment: Liver Function Change
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment switch. Treatment switching was defined as a prescription of another anticoagulant therapy that was started after treatment initiation of index anticoagulant treatment and within 30 days after estimated end of supply of index anticoagulant drug. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event. In this outcome measure, results for event "liver function change" are reported.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 1685 | 1446 | 352 | 306 | 230 | 1985 | 743
Participants
  Switched to Warfarin: Without Active Cancer: number analyzed (Participants) | 0 | 1155 | 76 | 104 | 71 | 867 | 120
  Switched to Warfarin: Without Active Cancer |  | 36 | 3 | 4 | 1 | 28 | 10
  Switched to NOAC: Without Active Cancer: number analyzed (Participants) | 1470 | 0 | 0 | 0 | 0 | 0 | 415
  Switched to NOAC: Without Active Cancer | 63 |  |  |  |  |  | 29
  Switched to PAC: Without Active Cancer: number analyzed (Participants) | 71 | 118 | 10 | 6 | 7 | 90 | 0
  Switched to PAC: Without Active Cancer | 7 | 11 | 0 | 1 | 0 | 10 |
  Switched to Apixaban: Without Active Cancer: number analyzed (Participants) | 118 | 0 | 0 | 38 | 42 | 334 | 68
  Switched to Apixaban: Without Active Cancer | 3 |  |  | 1 | 1 | 13 | 5
  Switched to Dabigatran: Without Active Cancer: number analyzed (Participants) | 141 | 0 | 17 | 0 | 16 | 130 | 48
  Switched to Dabigatran: Without Active Cancer | 6 |  | 0 |  | 2 | 4 | 4
  Switched to Edoxaban: Without Active Cancer: number analyzed (Participants) | 115 | 0 | 99 | 48 | 0 | 356 | 48
  Switched to Edoxaban: Without Active Cancer | 3 |  | 2 | 1 |  | 20 | 5
  Switched to Rivaroxaban: Without Active Cancer: number analyzed (Participants) | 1093 | 0 | 117 | 80 | 68 | 0 | 249
  Switched to Rivaroxaban: Without Active Cancer | 51 |  | 6 | 2 | 6 |  | 16
  Switched to Warfarin: With Active Cancer: number analyzed (Participants) | 0 | 84 | 5 | 10 | 3 | 64 | 36
  Switched to Warfarin: With Active Cancer |  | 3 | 1 | 0 | 0 | 2 | 1
  Switched to NOAC: With Active Cancer: number analyzed (Participants) | 98 | 0 | 0 | 0 | 0 | 0 | 172
  Switched to NOAC: With Active Cancer | 1 |  |  |  |  |  | 7
  Switched to PAC: With Active Cancer: number analyzed (Participants) | 46 | 89 | 5 | 4 | 7 | 73 | 0
  Switched to PAC: With Active Cancer | 3 | 0 | 0 | 0 | 0 | 0 |
  Switched to Apixaban: With Active Cancer: number analyzed (Participants) | 11 | 0 | 0 | 5 | 4 | 29 | 22
  Switched to Apixaban: With Active Cancer | 0 |  |  | 0 | 0 | 2 | 1
  Switched to Dabigatran: With Active Cancer: number analyzed (Participants) | 9 | 0 | 2 | 0 | 2 | 15 | 12
  Switched to Dabigatran: With Active Cancer | 0 |  | 0 |  | 0 | 0 | 0
  Switched to Edoxaban: With Active Cancer: number analyzed (Participants) | 6 | 0 | 7 | 1 | 0 | 27 | 23
  Switched to Edoxaban: With Active Cancer | 1 |  | 0 | 0 |  | 1 | 0
  Switched to Rivaroxaban: With Active Cancer: number analyzed (Participants) | 72 | 0 | 14 | 10 | 10 | 0 | 113
  Switched to Rivaroxaban: With Active Cancer | 0 |  | 0 | 0 | 1 |  | 6

18. Primary Outcome: Number of Participants With Clinical Events Preceding Index Anticoagulant Treatment Discontinuation
Description: Clinical event preceding first treatment change was defined as occurrence of any event (major bleeding, complications of VTE, thromboembolism, major surgeries, cancer-related event, kidney function change, liver function change) within 30 days before treatment discontinuation. Treatment discontinuation (complete discontinuation; no reinitiation) was defined as when a participant who ended their first continuous treatment episode with the index anticoagulant treatment without switching, and subsequently have no further prescriptions for that respective anticoagulant treatment during all available follow-up time. Index date was defined as date of first prescription for anticoagulants within 30 days after index VTE event.
Time Frame: Within 30 days before treatment discontinuation during observation period of maximum up to 88 months (retrospective data was retrieved and observed during 1 month of this study)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
Number analyzed (Participants) | 5151 | 22396 | 3107 | 1143 | 1311 | 16138 | 5983
Participants
  Major Bleeding: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Major Bleeding: Without Active Cancer | 42 | 118 | 13 | 7 | 5 | 90 | 20
  Complications of VTE: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Complications of VTE: Without Active Cancer | 10 | 25 | 4 | 2 | 3 | 15 | 18
  Thromboembolism: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Thromboembolism: Without Active Cancer | 258 | 777 | 123 | 48 | 53 | 537 | 734
  Major Surgery: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Major Surgery: Without Active Cancer | 78 | 1691 | 508 | 18 | 25 | 1138 | 625
  Cancer-related Event: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Cancer-related Event: Without Active Cancer | 133 | 307 | 40 | 14 | 20 | 232 | 291
  Kidney Function Changes: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Kidney Function Changes: Without Active Cancer | 104 | 240 | 39 | 13 | 11 | 172 | 383
  Liver Function Change: Without Active Cancer: number analyzed (Participants) | 4707 | 19826 | 2828 | 1028 | 1164 | 14170 | 4534
  Liver Function Change: Without Active Cancer | 158 | 452 | 65 | 34 | 28 | 321 | 441
  Major Bleeding: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Major Bleeding: With Active Cancer | 7 | 36 | 4 | 2 | 0 | 29 | 14
  Complications of VTE: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Complications of VTE: With Active Cancer | 1 | 2 | 0 | 0 | 0 | 2 | 0
  Thromboembolism: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Thromboembolism: With Active Cancer | 17 | 122 | 14 | 9 | 11 | 87 | 89
  Major Surgery: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Major Surgery: With Active Cancer | 11 | 66 | 7 | 1 | 5 | 52 | 190
  Cancer-related Event: With Active Cancer: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Kidney Function Changes: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Kidney Function Changes: With Active Cancer | 14 | 64 | 7 | 1 | 5 | 51 | 48
  Liver Function Change: With Active Cancer: number analyzed (Participants) | 444 | 2570 | 279 | 115 | 147 | 1968 | 1449
  Liver Function Change: With Active Cancer | 16 | 50 | 3 | 2 | 3 | 42 | 34

ADVERSE EVENTS:
Time Frame: Adverse events were not planned to be collected hence time frame was not applicable
Description: In this study individual participant data was not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (AE) cannot be met. Hence, AEs were not collected and reported in this study.
Arm/Group | Warfarin-Based Therapy | NOAC-Based Therapy: Apixaban | NOAC-Based Therapy: Dabigatran | NOAC-Based Therapy: Edoxaban | NOAC-Based Therapy: Rivaroxaban | PAC Only
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Phase 2 was not conducted due to insufficient statistical power that would lead to small and imbalanced sample sizes in comparison groups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT05022563/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/63/NCT05022563/SAP_001.pdf